CLINICAL TRIAL: NCT06986174
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Pacritinib in Relapsed or Refractory Waldenström Macroglobulinemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shayna Sarosiek, MD (Other)
Collaborators: Sobi, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Shayna Sarosiek, MD, Sponsor-Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-660
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Waldenström Macroglobulinemia; Lymphoplasmacytic Lymphoma; B-Cell Lymphoproliferative Disorder; Indolent Lymphoma
Keywords: Waldenström Macroglobulinemia; Lymphoplasmacytic Lymphoma; Lymphoma; B-Cell Lymphoproliferative Disorder; Indolent Lymphoma
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pacritinib (Experimental): 30 participants will complete:
  * Baseline visit with assessments and ECGs
  * Cycles 1 through 2 (28 days per cycle):
    --Day 1: Predetermined dose of Pacritinib 2x daily
  * Cycle 3, 6, 9, 12, and every 3 cycles for 48 cycles total (28 days per cycle):
    --Day 1: Predetermined dose of Pacritinib 2x daily
  * Bone marrow biopsies/aspirations at Cycles 6 and 12 and then yearly
  * End of Treatment visit with CT scan and bone marrow biopsy/aspiration
  * Follow up: every 12 weeks for 2 years
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Kinase inhibitor, capsule, taken orally per protocol.
  Other Names: SB1518; VONJO; Pacritinib Citrate

SUMMARY:
This study is being done to examine the safety and effectiveness of pacritinib as a possible treatment for participants with Waldenström macroglobulinemia (WM).

The name of the study drug involved in this study is:

-Pacritinib (a type of kinase inhibitor)

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase II study to evaluate the safety and efficacy of pacritinib in participants with symptomatic Waldenström macroglobulinemia (WM).

Pacritinib is a targeted therapy that blocks a protein called JAK2 that helps cells live and grow. It also inhibits IRAK1, which is important for the survival of WM cells. By blocking JAK2 & IRAK1, pacritinib may kill abnormal cells or stop them from growing.

The U.S. Food and Drug Administration (FDA) has not approved pacritinib for WM but it has been approved for Myelofibrosis.

The research study procedures include screening for eligibility, in-clinic visits, questionnaires, blood tests, urine tests, Computerized Tomography (CT) scans, X-rays, echocardiograms (ECGs), bone marrow biopsies and aspirations

Participants will receive study treatment for up to 4 years and will be followed for 2 years, or until there is start of a new treatment.

It is expected that about 30 people will take part in this research study.

Sobi AG, Inc. is supporting this research study by providing study drug and funding.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ECOG performance status ≤2
* Clinicopathological diagnosis of Waldenström Macroglobulinemia
* Symptomatic disease meeting criteria for treatment using consensus panel criteria from the Second International Workshop on Waldenström macroglobulinemia. At least one of the following:

  * constitutional symptoms: recurrent fever, night sweats, fatigue or weight loss
  * progressive or symptomatic lymphadenopathy or splenomegaly
  * hemoglobin ≤10 g/dL
  * platelet count ≤100 k/uL
  * hyperviscosity syndrome
  * symptomatic peripheral neuropathy
  * systemic amyloidosis
  * renal insufficiency
  * symptomatic cryoglobulinemia
* Serum IgM level ≥ 2 times the upper limit of normal
* Participants must meet the following organ and marrow functions as defined below:

  * absolute neutrophil count ≥0.5 k/uL without growth factor within 7 days
  * platelet count ≥50 k/uL without platelet transfusion within 7 days
  * total bilirubin ≤1.5 times the upper limit of normal or ≤3 times the upper limit of normal with documented liver involvement, hemolysis or Gilbert's disease
  * AST (SGOT) and ALT (SGPT) ≤2.5 times the upper limit of normal or ≤5 times the upper limit of normal with documented liver involvement
  * Creatinine clearance ≥30 ml/min using Cockcroft/Gault equation
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)
* At least 2 prior lines of treatment for Waldenström Macroglobulinemia. Participants must either be BTK inhibitor exposed or not be a candidate for BTK therapy.
* Women of childbearing potential: Females of childbearing potential (FCBP) will be required to use two highly effective forms of contraception simultaneously or will remain abstinent from heterosexual intercourse during the following periods related to this study:

  1. while participating in the study; and 2) for at least three months (90 days) after discontinuation from the study. FCBP must be referred to a qualified provider of contraceptive methods if needed.

Exclusion Criteria:

* Current history of uncontrolled HIV
* Patients with a known history of HIV must have a viral load assessed for eligibility and must be on a stable antiretroviral regimen that can be administered concurrent with pacritinib.
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection based on criteria below

  * Hepatitis B virus (HBV): Patients with positive hepatitis B surface antigen (HBsAg) are excluded. Patients with positive hepatitis B core antibody (antiHBc) and negative HBsAg require hepatitis B polymerase chain reaction (PCR) evaluation before enrollment. Patients who are hepatitis B PCR positive will be excluded.
  * Hepatitis C virus (HCV): positive hepatitis C antibody. If positive hepatitis C antibody result, patient will need to have a negative result for hepatitis C ribonucleic acid (RNA) before enrollment. Patients who are hepatitis C RNA positive will be excluded.
* Participants with chronic liver disease and hepatic impairment meeting Child-Pugh class B or C (Appendix B)
* Participants who are pregnant, breast feeding, or planning to become pregnant while enrolled in this study or within 3 month after last study dose (2 weeks for breastfeeding)
* Current CNS involvement by WM
* Active alcohol or drug abuse
* Concurrent administration of medications that are moderate or strong inhibitors or inducers of CYP3A within 14 days or 5 half-lives, whichever is shorter, prior to first dose of study drug.
* Concurrent participation in another therapeutic clinical trial
* History of another malignancy, except adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, localized prostate cancer, or other adequately treated cancer currently in complete remission
* Prior or ongoing clinically significant illness, including active infections requiring antibiotics, of medical condition that, in the investigator's opinion, could affect the safety of the patient; alter the absorption, distribution, metabolism or excretion of the study drug; or impair the assessment of study results
* Inability to swallow pills
* Significant cardiovascular disease defined as:

  * Unstable angina, or
  * History of myocardial infarction within 6 months prior to planned start
  * Previously documented left ventricular ejection fraction (LVEF) by any method of ≤ 45% in the 12 months prior to planned start; assessment of LVEF via echocardiogram or multigated acquisition (MUGA) scan during screening should be performed in selected patients as medically indicated, or
  * Any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or
  * Uncontrolled or symptomatic arrhythmias
* Prolonged QT Interval with baseline QTc >480 msec using the Bazette formula
* Ongoing, active infection.
* Active bleeding requiring blood transfusion or other medical intervention. Participants requiring anticoagulation therapy are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 48 months
  ORR was defined as the percentage of participants achieving complete response (CR), very good partial response (VGPR), partial response (PR) and minimal response (MR) on treatment based on IWWM-11 criteria.

SECONDARY OUTCOMES:
Complete Response Rate | Up to 48 months
  Complete response rate was defined as the percentage of participants achieving complete response (CR) on treatment based on IWWM-11 criteria, defined as having resolution of WM related symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, and resolution of any adenopathy or splenomegaly. A complete response requires reconfirmation demonstrating normal serum IgM levels, and absence of IgM paraprotein by immunofixation by a measurement repeated at least 2 weeks later.
Very Good Partial Response Rate | Up to 48 months
  Very good partial response rate was defined as the percentage of participants achieving very good partial response (VGPR) on treatment based on IWWM-11 criteria, defined as ≥90% reduction in serum IgM levels, or normalization of serum IgM levels with persistent IgM monoclonal spike in SPEP or immunofixation.
Partial Response Rate | Up to 48 months
  Partial response rate was defined as the percentage of participants achieving partial response (PR) on treatment based on IWWM-11 criteria, Partial response (PR) is defined as achieving a ≥50% to <90% reduction in serum IgM levels.
Minimal Response Rate | Up to 48 months
  Minimal response rate was defined as the percentage of participants achieving minimal response (MR) on treatment based on IWWM-11 criteria, defined as ≥25 to <50% reduction in serum IgM levels.
Stable Disease Rate | Up to 48 months
  Stable disease rate was defined as the percentage of participants achieving stable disease (SD) on treatment based on IWWM-11 criteria, defined as <25% reduction to <25% increase in serum IgM levels.
Progressive Disease Rate | Up to 48 months
  Stable disease rate was defined as the percentage of participants achieving progressive disease (SD) on treatment based on IWWM-11 criteria, defined as defined as a≥25% increase in serum IgM level occurring with an absolute increase of at least 500 mg/dL from nadir or progression of clinically significant disease-related symptom(s). Reconfirmation of the initial IgM increase is required when IgM is the sole criterion for progressive disease confirmation. Death from any cause or initiation of a new anti-neoplastic therapy will also be considered a progression event. Additionally, a new lesion (>1.5 cm in any axis) or unequivocal evidence of an increase by >50% in any axis to >1.5 cm in size of previously involved extramedullary disease sites from their nadir measurement. Development of Bing Neel syndrome, amyloidosis, or other extramedullary disease manifestations, as well as disease transformation will be considered as progressive events.
Time to Response (TTR) | Up to 48 months
  TTR is the time from treatment initiation until the attainment of a minor response.
Time to Major Response (TTMR) | Up to 48 months
  TTMR is the time from treatment initiation until attaining a PR or better.
Median Progression-free Survival (PFS) | Up to 48 months
  PFS based on Kaplan-Meier methodology is defined as the time from treatment initiation until disease progression, death from any cause, or last follow-up visit.
Time to Next Treatment (TTNT) | Up to 48 months
  TTNT is the time between treatment initiation and initiation of the next therapy.
Median Overall Survival (OS) | Up to 6 years
  OS is defined as the time from treatment initiation until death from any cause or last follow-up visit
Bone marrow response | Up to 48 months
  Absolute change in bone marrow burden of disease from baseline
Overall Response Rate Among Participants Without MYD88 Mutations | Up to 48 months
  Overall Response Rate in participants who tested negative for a MYD88 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants With MYD88 Mutations | Up to 48 months
  Overall Response Rate in participants who tested positive for a MYD88 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants Without CXCR4 Mutations | Up to 48 months
  Overall Response Rate in participants who tested negative for a CXCR4 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants With CXCR4 Mutations | Up to 48 months
  Overall Response Rate in participants who tested positive for a CXCR4 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants With TP53 Mutations | Up to 48 months
  Overall Response Rate in participants who tested positive for a TP53 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Overall Response Rate Among Participants Without TP53 Mutations | Up to 48 months
  Overall Response Rate in participants who tested negative for a TP53 mutation= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).
Number of Participants With Treatment-related Adverse Events | Up to 48 months
  Number of participants who experienced an adverse event while on pacritinib
Overall Response Rate Among Participants who progressed on covalent BTK-inhibitors | Up to 48 months
  Overall Response Rate in participants who previously progressed on covalent BTK inhibitors= Minor response (>25%-50% reduction in serum IgM from baseline) + Partial Response (>50-90% reduction in serum IgM from baseline) + Very Good Partial Response (>90% reduction in serum IgM from baseline) + Complete Response (resolution of all symptoms, normalization of serum IgM with disappearance of IgM paraprotein, resolution of any adenopathy or splenomegaly).

CONTACTS AND LOCATIONS:
Overall Officials: Shayna Sarosiek, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu